CLINICAL TRIAL: NCT03023150
Title: Ischemic Preconditioning as an Intervention to Improve Stroke Rehabilitation
Brief Title: Ischemic Preconditioning as an Intervention to Improve Stroke Rehabilitation - Froedtert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Matthew J. Durand, Assistant Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRO00027450
Record Dates: First submitted 2017-01-03; First posted 2017-01-18 (Estimated); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Stroke Rehabilitation; Ischemic Preconditioning; Physical and Rehabilitation Medicine
MeSH Terms: interventions — Ischemic Preconditioning; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ischemic Preconditioning (Experimental): Inflation of blood pressure cuff to 225 mmHg on paretic leg. 1 session: 5 minutes of inflation, 5 minutes deflation, repeated 5 times.
  Interventions: Other: Ischemic Preconditioning
- Sham (Sham Comparator): Inflation of blood pressure cuff to 25 mmHg on paretic leg. 1 session: 5 minutes of inflation, 5 minutes deflation, repeated 5 times.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Ischemic Preconditioning
  Arms: Ischemic Preconditioning
Other: Sham
  Arms: Sham

SUMMARY:
This study will be the first study to use ischemic preconditioning (IPC) as an intervention to improve stroke rehabilitation. IPC is a well studied, well tolerated intervention which has been shown to improve regional blood flow, motor neuron excitability and muscle function in multiple patient groups and in young, healthy subjects. Because IPC targets three physiological systems which are all affected by stroke, we hypothesize that repeated bouts of IPC during the first days to months following stroke (when the majority of recovery occurs) will make traditional rehabilitation strategies more effective.

ELIGIBILITY:
Inclusion Criteria:

1. be between the ages of 40-80
2. able to give informed consent.
3. be < 6 months post diagnosis of unilateral cortical stroke and
4. have residual leg paresis.

Exclusion Criteria:

1. chronic low back or hip pain
2. substance abuse
3. head trauma with loss of conciousness in last 6 months
4. neurodegenerative disorder
5. participant taking any medication or supplement that adversely interacts with nitroglycerin (exclusion from nitro administration only, applies to outpatients only)
6. participant has a known allergy to nitroglycerin (exclusion from nitro administration only, applies to outpatients only)
7. resting systolic blood pressure < 90mmHg (exclusion from nitro administration only, applies to outpatients only)
8. any condition where knee extension contractions are contraindicated
9. people who are unable to follow multi step commands.
10. pregnancy (DXA scan exclusion only)
11. history of major psychiatric disorder
12. participant has had a myocardial infarction in the last year
13. participant has stage II hypertension (BP>160/100)
14. participant is unable to contract knee muscles
15. participant is unable to sit upright for 2 hours
16. participant has a resting heart rate >100 beats per minute
17. history of multiple strokes

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10; Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
Change in Knee Extensor Strength | Admission into study and within 3 days of Discharge from Froedtert Hospital

SECONDARY OUTCOMES:
Change in Walking Speed | Admission into study and within 3 days of Discharge from Froedtert Hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Undecided